CLINICAL TRIAL: NCT04356911
Title: The Association of Strontium Chloride With Photobiomodulation in the Control of Tooth Post-bleaching Sensitivity: Clinical Trial, Randomized, Double-blind and Split-mouth.
Brief Title: The Strontium Chloride Associated With Photobiomodulation in the Control of Post-bleaching Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Cecy Martins Silva, Associate Professor, Universidade Federal do Para
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-007
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PLACEBO (Negative Control) (Placebo Comparator): The dental elements of this group had no desensitizing treatment. After whitening therapy, a water-soluble placebo gel (KY®, Johnson & Johnson, SP, Brazil) was applied to dental oral surfaces, then the laser tip was positioned at two points, apical and cervical, without emitting light (placebo), simulating the application of Low Level Laser Therapy (LLLT).
  Interventions: Other: PLACEBO (Negative Control)
- FBM (Experimental): The group received the application of a placebo gel associated with LLLT after office bleaching.
  Interventions: Other: FBM
- ESTRÔNCIO (Experimental): After whitening in-office bleaching, the group was treated with desensitization to 10% strontium chloride. Subsequently, a laser tip was positioned at two points (apical and cervical), without emitting light (placebo).
  Interventions: Other: ESTRÔNCIO
- FBM+ESTRÔNCIO (Experimental): After whitening in the office, the group received a 10% strontium chloride desensitizer associated with low level light therapy.
  Interventions: Other: FBM+ESTRÔNCIO

INTERVENTIONS:
Other: PLACEBO (Negative Control) — The group received in-office bleaching. A 45-minute application of 35% hydrogen peroxide gel (Whiteness HP, FGM, Joinville, SC) was carried. After whitening therapy, a water-soluble placebo gel (KY®, Johnson & Johnson, SP, Brazil) was applied to the buccal surfaces of incisors, canines and premolars with the help of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo , Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a handpiece at low speed (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to rub the placebo gel for 20 seconds in each tooth surface. After washing the placebo gel, the laser tip was positioned at two points, apical and cervical, without emitting light (placebo), simulating the application of low-level laser therapy (LLLT).
  This protocol was performed in 3 sessions, with an interval of seven days between them.
  Arms: PLACEBO (Negative Control)
Other: FBM — This group received photobimodulation with low level laser therapy (LLLT) of infrared spectrum with a wavelength of 808 nm in its active environment AsGaAl (Photon Lase III, DMC Equipamentos Ltda; São Carlos, SP, Brazil), at two points: cervical and apical region of the incisors, canines and premolars. 60 J / cm² was applied at each point for 16 seconds. The laser was applied in 3 sessions with a time interval of seven days between them.
  Arms: FBM
Other: ESTRÔNCIO — After whitening therapy, a toothpaste with 10% strontium chloride (Sensodyne Original, GSK, London, United Kingdom) was applied to the buccal surfaces of incisors, canines and premolars with the help of a Microbrush applicator (Microbrush, 3M ESPE, São Paulo , Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a handpiece at low speed (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to rub the desensitizer for 20 seconds on each tooth , according to the manufacturer's specifications. The desensitizer therapy was realized in 3 sessions with a time interval of seven days between them.
  Arms: ESTRÔNCIO
Other: FBM+ESTRÔNCIO — After whitening therapy, a 10% strontium chloride toothpaste (Sensodyne Original, GSK, London, United Kingdom) was applied to the buccal surfaces of whitened teeth with the help of a Microbrush applicator applicator (Microbrush, 3M ESPE, São Paulo , Brazil) for 10 minutes. Then, a rubber cup (Unid Microdont, São Paulo, SP, Brazil) mounted on a handpiece at low speed (Dabi Atlante, Ribeirão Preto, SO, Brazil) was used to rub the desensitizer for 20 seconds on each tooth , according to the manufacturer's specifications. After washing the desensitizer, the photobimodulation was realized with Low Level Laser Therapy (LLLT) of infrared spectrum with wavelength of 808 nm in its active environment AsGaAl (Photon Lase III, DMC Equipamentos Ltda; São Carlos, SP, Brazil), in two points: cervical and apical region of the incisors, canines and premolars. 60 J / cm² was applied at each point for 16 seconds. This protocol was performed in 3 sessions, with an interval of seven days between them.
  Arms: FBM+ESTRÔNCIO

SUMMARY:
This study investigated the effects of the association of strontium chloride with photobiomodulation on the dental bleaching process, testing the hypothesis that they may control dental sensitivity post-bleaching teeth.

DETAILED DESCRIPTION:
The objective of this double-blind, randomized, controlled clinical study was to evaluate the effect of 10% strontium chloride associated with photobiomodulation (FBM) on teeth exposed to 35% hydrogen peroxide during 3 weeks of whitening treatment. Methods: 50 volunteers were evaluated by the split mouth model, where the hemiarchy patients were randomized and subsequently allocated to one of the experimental groups: PLACEBO (negative control) - group with no desensitizing treatment, only bleached; FBM (positive control) - group treated with placebo gel and application of the LLLT (Low Level Laser Therapy); ESTRÔNCIO (positive control) - group treated with 10% strontium chloride and simulation of LLLT application (without light emission); and FBM + ESTRÔNCIO - group treated with LLLT + 10% strontium chloride.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* absence of active caries lesions
* never having undergone previous whitening therapy
* not present dental hypersensitivity
* don't be a smoker
* not be pregnant
* present at least 28 teeth in the oral cavity.

Exclusion Criteria:

* volunteers who were under orthodontic treatment,
* presence of periodontal disease
* dental cracks or fractures
* restorations and prostheses on anterior teeth
* extensive molar restorations
* gastroesophageal disorders
* severe internal dental darkening
* presence of dentinal exposure in anterior and / or posterior teeth.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of desensitizer treatment in the control of tooth post-bleaching sensitivity (P21) | 21 days
  Self-reported pain intensity was assessed daily, during 21 days, through self-perception questionnaire, answered by the patients from the first tooth bleaching session until one week after the last session. The evaluation was performed by each patient, according to a modified visual analog scale, as follows: 0- no pain, 1 mild pain, 2 - moderate pain and 3 -severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, PhD, Principal Investigator — clinical professor
Locations (1):
- Para's Federal University, Belém, Pará, Brazil